CLINICAL TRIAL: NCT03400904
Title: Gestion du Sevrage de la Ventilation mécanique du Patient neurolésé en réanimation et Association Avec le Devenir. Etude Observationnelle Multi-centrique Internationale. Extubation Strategies in Neuro-Intensive Care Unit Patients and Associations With Outcome. The International Observational ENIO Study.
Brief Title: Extubation Strategies in Neuro-Intensive Care Unit Patients and Associations With Outcome.
Acronym: ENIO
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0328
Record Dates: First submitted 2018-01-02; First posted 2018-01-17 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries | interventions — Tracheostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with brain injury and mechanical ventilation exposed to extubation/tracheostomy — Extubation and/or tracheostomy if applicable

SUMMARY:
Rationale Prolonged mechanical ventilation (MV) is common in patients with severe Brain Injury (BI). Guidelines for the management of extubation are largely lacking for patients with BI, and the role of tracheostomy is highly uncertain. More important, data on practice of management of extubation is yet underreported, as is the use of tracheotomy in this specific subset of critical care patients.

Objective The objective of this prospective observational study is to describe the management of extubation and tracheostomy in intensive care unit (ICU) patients with BI. The aim is to describe the incidence of extubation failure and the rate of tracheostomy.

Study design The "Extubation strategies in Neuro-Intensive care unit patients, and associations with Outcomes (ENIO)" is an observational multicentre international cohort study.

Study population The investigators will include patients undergoing BI, with an initial Glasgow Coma Score ≤ 12 and with a delivered duration of mechanical ventilation (MV) ≥ 24 hours at ICU admission. The inclusion period will last 6 months in total, and each centre is expected to include at least 24 patients during this period. With over 60 ICUs participating worldwide, we expect to include 1500 patients.

Main parameters Parameters to be collected include: general neurological management, ventilatory management, general ICU complications, specific data on extubation and tracheostomy, general in-ICU outcomes and in-hospital mortality.

Nature and extent of the burden and risks associated with participation Because of the observational design of the study using routinely collected data, there is no additional burden for the patient. Collection of data from ICU charts and/or (written or electronic) medical records systems bears no risk to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years' old
* Patients admitted in a ICU for a central neurological pathology, listed as follows, with estimated or clinically evaluated Glasgow Coma Score ≤12 before endo-tracheal intubation, with anomaly on brain CT-scan and requiring effective invasive mechanical ventilation ≥ 24 hours are eligible to the study:
* Traumatic Brain Injury
* Aneurysmal Subarachnoid haemorrhage
* Intra-Cranial Haemorrhage
* Ischemic Stroke
* Central Nervous System Infection (Abscess, Empyema, Meningitides, Encephalitis…)
* Brain Tumour
* Patient with an attempt of extubation and/or performance of a tracheostomy

Exclusion Criteria:

* Patients < 18 years' old
* Patients with ongoing pregnancy
* Patients with spine cord injury above T4
* Resuscitated cardiac arrest
* Withdrawal of Life-Sustaining Treatment (WLST) in the first 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing significant brain injury, with a mechanical ventilation duration≥ 24 hours and baseline Gasgow coma score ≤12, undergoing an attempt of extubation and/or tracheostomy
Sampling Method: Non-Probability Sample
Enrollment: 1750 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Extubation success | Extubation failure will be defined as the need to re-intubate the patient within 48hours after removal
  Successful removal of endo-tracheal tube
Extubation success | Extubation failure will be defined as the need to re-intubate the patient within 96hours after removal
  Successful removal of endo-tracheal tube
Extubation success | Extubation failure will be defined as the need to re-intubate the patient within 168hours (7 days) after removal
  Successful removal of endo-tracheal tube

SECONDARY OUTCOMES:
In-ICU VAP | Onset of VAP during ICU stay and after extubation failure, when appropriate (Median 15 days)
  Ventilator-acquired pneumonia (VAP)
Mechanical ventilation duration | ICU-stay (Median 15 days)
  Calculation of the duration of Mechanical Ventilation during ICU stay.
Tracheostomy | ICU stay (Median 15 days)
  Study the rate and reasons for tracheostomy in patients with brain injury
In-ICU mortality | During ICU stay (Median 15 days)
  Death in the ICU
In-hopsital mortality | During the first hospital stay following Brain-Injury (Median 25 days)
  Death during hospitalization

CONTACTS AND LOCATIONS:
Locations (6):
- Nantes University Hospital, Nantes, France
- Varanasi BHU Hospital, Varanasi, India
- University of Genes, Genova, Italy
- Netherlands (3):
  - University of Amsterdam, Amsterdam
  - Enschede (Medisch Spectrum Twente), Enschede
  - Haaglanden (Medical Center), The Hague

IPD SHARING:
Plan to Share IPD: Yes
All proposals for sub-studies on the main ENIO database are encouraged. Secondary studies must be approved by the steering committee. Study results will be presented and disseminated in a timely manner. Authorship will be proposed by the investigators of the sub-studies and approved by the steering committee. National groups may enter requests for data-access to analyse their national datasets. Owing to the full anonymization of data according to European Union laws and regulations, institutional datasets will not be available.
Time Frame: No time limit

REFERENCES:
- [Derived] Daza JF, Hamad DM, Urner M, Liu K, Wahlster S, Robba C, Stevens RD, McCredie VA, Cinotti R, Taran S; ENIO Study Group; PROtective VENTilation Network; European Society of Intensive Care Medicine; Colegio Mexicano de Medicina Critica; AtlanRea Group; Societe Francaise d'Anesthesie-Reanimation-SFAR Research Network. Low-Tidal-Volume Ventilation and Mortality in Patients With Acute Brain Injury: A Secondary Analysis of an International Observational Study. Chest. 2025 Nov;168(5):1141-1151. doi: 10.1016/j.chest.2025.06.042. Epub 2025 Jul 8. PMID 40639639
- [Derived] van Vliet R, van Meenen DMP, Robba C, Cinotti R, Asehnoune K, Stevens RD, Battaglini D, Taran S, van der Jagt M, Taccone FS, Paulus F, Schultz MJ; ENIO investigators. Association of age with extubation failure in neurocritical intensive care unit patients--Insight from an international prospective study named ENIO. J Crit Care. 2025 Aug;88:155067. doi: 10.1016/j.jcrc.2025.155067. Epub 2025 Apr 3. PMID 40184992
- [Derived] Serafini SC, Cinotti R, Asehnoune K, Battaglini D, Robba C, Neto AS, Pisani L, Mazzinari G, Tschernko EM, Schultz MJ; PRoVENT, the PRoVENT-iMiC and ENIO, investigators. Potentially modifiable ventilation factors associated with outcome in neurocritical care vs. non-neurocritical care patients: Rational and protocol for a patient-level analysis of PRoVENT, PRoVENT-iMiC and ENIO (PRIME). Rev Esp Anestesiol Reanim (Engl Ed). 2025 May;72(5):501690. doi: 10.1016/j.redare.2025.501690. Epub 2025 Feb 15. PMID 39961531
- [Derived] Taran S, Perrot B, Angriman F, Cinotti R; Extubation strategies in Neuro-Intensive care unit patients and associations with Outcomes (ENIO) Study Group; PROtective VENTilation network; European Society of Intensive Care Medicine; Colegio Mexicano de Medicina Critica; Atlanrea group, and the Societe Francaise d'Anesthesie et de Reanimation (SFAR) research network; Extubation strategies in Neuro-Intensive care unit patients and associations with Outcomes (ENIO) Study Group and PROtective VENTilation network and the European Society of Intensive Care Medicine and the Colegio Mexicano de Medicina Critica and the Atlanrea group, and the Societe Francaise d'Anesthesie et de Reanimation (SFAR) research network. Evaluating the Sum of Eye and Motor Components of the Glasgow Coma Score As a Predictor of Extubation Failure in Patients With Acute Brain Injury. Crit Care Med. 2024 Aug 1;52(8):1258-1263. doi: 10.1097/CCM.0000000000006283. Epub 2024 Apr 1. PMID 38557684
- [Derived] Taran S, Diaz-Cruz C, Perrot B, Alvarez P, Godoy DA, Gurjar M, Haenggi M, Mijangos JC, Pelosi P, Robba C, Schultz MJ, Ueno Y, Asehnoune K, Cho SM, Yarnell CJ, Cinotti R, Stevens RD. Association of Noninvasive Respiratory Support with Extubation Outcomes in Brain-injured Patients Receiving Mechanical Ventilation: A Secondary Analysis of the ENIO Prospective Observational Study. Am J Respir Crit Care Med. 2023 Aug 1;208(3):270-279. doi: 10.1164/rccm.202212-2249OC. PMID 37192445
- [Derived] Wahlster S, Sharma M, Taran S, Town JA, Stevens RD, Cinotti R, Asehoune K, Pelosi P, Robba C; ENIO Study Group Collaborators. Utilization of mechanical power and associations with clinical outcomes in brain injured patients: a secondary analysis of the extubation strategies in neuro-intensive care unit patients and associations with outcome (ENIO) trial. Crit Care. 2023 Apr 20;27(1):156. doi: 10.1186/s13054-023-04410-z. PMID 37081474
- [Derived] Cinotti R, Pelosi P, Schultz MJ, Aikaterini I, Alvarez P, Badenes R, Mc Credie V, Elbuzidi AS, Elhadi M, Godoy DA, Gurjar M, Haenggi M, Kaye C, Mijangos-Mendez JC, Piagnerelli M, Piracchio R, Reza ST, Stevens RD, Yoshitoyo U, Asehnoune K; ENIO Study Group. Extubation strategies in neuro-intensive care unit patients and associations with outcomes: the ENIO multicentre international observational study. Ann Transl Med. 2020 Apr;8(7):503. doi: 10.21037/atm.2020.03.160. PMID 32395547